CLINICAL TRIAL: NCT04758338
Title: Enhancing Cancer Care Of Rural Dwellers Through Telehealth and Engagement (ENCORE)
Brief Title: Enhancing Cancer Care Of Rural Dwellers
Acronym: ENCORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debra Friedman (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Debra Friedman, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC PED 2013; R01CA240093-01 (NIH)
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTS Program Arm (Experimental): 6-week intervention delivered via telehealth using the VUMC telehealth services.
  Interventions: Other: VUMC telehealth services; Other: Interview
- Education Attention Control Arm (Active Comparator): Receive educational materials either online, by email, or in print form.
  Interventions: Other: Educational materials

INTERVENTIONS:
Other: VUMC telehealth services — Participants will access the CTS link (sent to them via email), which will connect them directly to a videoconference and enable them to see and hear the facilitators and other patients in the group.
  Arms: CTS Program Arm
Other: Interview — 25-30 participants will be interviewed
  Arms: CTS Program Arm
Other: Educational materials — Participants will be provided educational materials
  Arms: Education Attention Control Arm

SUMMARY:
Through a multi-level remote intervention, the Vanderbilt-Ingram Cancer Center (VICC) seeks to improve comprehensive cancer care delivery to patients residing in rural communities with persistent poverty. We plan to do this by using telehealth to broaden the reach of our NCI-designated comprehensive cancer center in these communities

DETAILED DESCRIPTION:
Objectives:

* Evaluate the clinical effectiveness of a multi-level telehealth-based intervention for rural hospitals consisting of provider access to tumor board expertise that incorporates disease, patient and molecular tumor characteristics, together with patient access to a supportive care intervention to improve cancer care delivery.
* Evaluate the facilitators and barriers to future larger-scale dissemination and implementation of the multi-level intervention, designed to enhance quality rural cancer care delivery.

ELIGIBILITY:
Inclusion Criteria:

Provider and Patient:

- At least 21 years of age or older and English speaking with the ability to provide informed consent

* Oncology providers within designated VHAN oncology practices
* Newly diagnosed or relapsed cancer patients of aforementioned oncology providers

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Measure the effectiveness of a multi-level telehealth-based intervention | Approximately 3 years
Estimate the facilitators to a future large-scale multi-level intervention | Approximately 3 years
Estimate the barriers to a future large-scale multi-level intervention | Approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (5):
- United States (5):
  - Baptist Cancer Center- Golden Triangle Columbus, Columbus, Mississippi
  - Baptist Cancer Center - North Mississippi, Oxford, Mississippi
  - Baptist Cancer Center- Bartlett, Bartlett, Tennessee
  - Ballad Health Systems, Kingsport, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pal T, Hull PC, Koyama T, Lammers P, Martinez D, McArthy J, Schremp E, Tezak A, Washburn A, Whisenant JG, Friedman DL. Enhancing Cancer care of rural dwellers through telehealth and engagement (ENCORE): protocol to evaluate effectiveness of a multi-level telehealth-based intervention to improve rural cancer care delivery. BMC Cancer. 2021 Nov 23;21(1):1262. doi: 10.1186/s12885-021-08949-4. PMID 34814868

DOCUMENTS (1):
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT04758338/ICF_000.pdf